CLINICAL TRIAL: NCT03333343
Title: A Phase Ib, Open Label, Multi-center Study to Characterize the Safety, Tolerability and Preliminary Efficacy of EGF816 in Combination With Selected Targeted Agents in EGFR Mutant NSCLC
Brief Title: Study of EGF816 in Combination With Selected Targeted Agents in EGFR-mutant NSCLC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEGF816X2102; 2024-511757-21-00 (Other: CTIS Number)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: EGFR-mutant Non-small Cell Lung Cancer
Keywords: EGFR-mutant NSCLC; EGF816; LXH254; INC280; ribociclib; trametinib; gefitinib; EGFR T790M; BRAF mutation; BRAF fusion; BRAF rearrangement; MET amplification
MeSH Terms: interventions — nazartinib; trametinib; ribociclib; naporafenib; capmatinib; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Arm 1 (Experimental): EGF816+ trametinib in escalation phase
  Interventions: Drug: EGF816; Drug: trametinib
- Arm 2 (Experimental): EGF816 + ribociclib in escalation phase
  Interventions: Drug: EGF816; Drug: ribociclib
- Arm 3 (Experimental): EGF816 + LXH254 in escalation phase
  Interventions: Drug: EGF816; Drug: LXH254
- Arm A (Experimental): EGF816 + INC280 in expansion phase (patients with no known resistance mechanism)
  Interventions: Drug: EGF816; Drug: INC280
- Arm B (Experimental): EGF816 + trametinib in expansion phase
  Interventions: Drug: EGF816; Drug: trametinib
- Arm C (Experimental): EGF816 + ribociclib in expansion phase
  Interventions: Drug: EGF816; Drug: ribociclib
- Arm D (Experimental): EGF816 + LXH254 in expansion phase (patients with no known resistance mechanism)
  Interventions: Drug: EGF816; Drug: LXH254
- Arm E (Experimental): EGF816 + LXH254 in expansion phase (patients with known resistance mechanism)
  Interventions: Drug: EGF816; Drug: LXH254
- Arm F (Experimental): EGF816 + gefitinib in expansion phase
  Interventions: Drug: EGF816; Drug: gefitinib
- Arm G (Experimental): EGF816 + INC280 in expansion phase (patients with known resistance mechanism)
  Interventions: Drug: EGF816; Drug: INC280

INTERVENTIONS:
Drug: EGF816 — Study Drug
Drug: trametinib — Study Drug
  Arms: Arm 1; Arm B
Drug: ribociclib — Study Drug
  Arms: Arm 2; Arm C
Drug: LXH254 — Study Drug
  Arms: Arm 3; Arm D; Arm E
Drug: INC280 — Study Drug
  Arms: Arm A; Arm G
Drug: gefitinib — Study Drug
  Arms: Arm F

SUMMARY:
The study purpose is to evaluate the safety, tolerability, and preliminary efficacy of the addition of INC280, trametinib, ribociclib, gefitinib, or LXH254 to EGF816 in adult patients with advanced Epidermal growth factor receptor- mutant (EGFR-mutant) non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase Ib, open label, non-randomized dose escalation study of EGF816 in combination with ribociclib, trametinib, or LXH254, followed by dose expansion of EGF816 in combination with ribociclib, trametinib, LXH254, INC280, or gefitinib in adult patients with advanced EGFR-mutant NSCLC.

During the dose escalation part, patients were assigned to the addition of trametinib, ribociclib, or LXH254 to EGF816.

Following determination of the recommended dose for the combination of EGF816 + trametinib, EGF816 + ribociclib, and EGF816 + LXH254, patients could be enrolled to the dose expansion arms of each of these combinations. Patients could also be assigned to EGF816 + INC280. The planned arm EGF816 + gefitinib in dose expansion was not opened for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed locally advanced (stage IIIB) or metastatic (stage IV) EGFR mutant (ex19del, L858R) NSCLC.
* Requirements of EGFR mutation status and prior lines of treatment:
* Treatment naive patients, who have locally advanced or metastatic NSCLC with EGFR sensitizing mutation (e.g., L858R and/or ex19del), have not received any systemic antineoplastic therapy for advanced NSCLC and are eligible to receive EGFR TKI treatment. Patients with EGFR exon 20 insertion/duplication are not eligible. Note: patients who have received only one cycle of chemotherapy in the advanced setting are allowed.
* Patients who have locally advanced or metastatic NSCLC with EGFR sensitizing mutation AND an acquired T790M mutation (e.g., L858R and/or ex19del, T790M+) following progression on prior treatment with a 1st-generation EGFR TKI or 2nd-generation EGFR TKI. These patients may not have received more than 4 prior lines of antineoplastic therapy in the advanced setting, including EGFR TKI, and may not have received any agent targeting EGFR T790M mutation (i.e., 3rd-generation EGFR TKI).
* Patients who have locally advanced or metastatic NSCLC with EGFR sensitizing mutation and a "de novo" T790M mutation (i.e., no prior treatment with any agent known to inhibit EGFR including EGFR TKI). These patients may not have received more than 3 prior lines of antineoplastic therapy in the advanced setting, and may not have received any prior 3rd generation EGFR TKI.
* Patients must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patients must be willing to undergo a new tumor biopsy during therapy on this study, and at screening if an archival tumor sample obtained since the diagnosis of advanced disease (1L patients) or since last treatment failure (2L+ patients) is not available.

Exclusion Criteria:

* Patients with a history or presence of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis.
* Patients with unstable brain metastases.
* Patients with a history of another malignancy.
* Patients with a known history of human immunodeficiency virus (HIV) seropositivity.
* Patients with clinically significant, uncontrolled heart disease.
* Patients participating in additional parallel investigational drug or medical device studies.
* Prior therapies:
* Patients who have been treated with EGFR TKI in the adjuvant setting within 6 months, unless acquired EGFR T790M is present in a tumor or blood sample obtained since the discontinuation of the EGFR TKI.
* Patients who have been treated with prior EGFR TKI targeting T790M (3rd generation).
* Patients who have been treated with systemic anti-neoplastic therapy within:

  * 2 weeks for fluoropyrimidine monotherapy
  * 6 weeks for nitrosoureas and mitomycin
  * 4 weeks or ≤ 5 half-lives (whichever is shorter) for biological therapy (including monoclonal antibodies) and continuous or intermittent small molecule therapeutics or any other investigational agent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events and serious adverse events | Every day until study end, approximately 4 years
  Assess safety and tolerability including incidence of dose limiting toxicities, adverse events, and serious adverse events.
Number of participants with DLTs in the first cycle of combination (Dose escalation only) | 28 days
  A Dose-Limiting Toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications that occurs within the first 28 days of combination treatment during the dose escalation part of the study. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Number of participants with dose interruptions and reductions | From first dose until study ends, approximately 4 years
  Assessment of tolerability. For patients who do not tolerate the protocol-specified dosing schedule, dose adjustments may be permitted in order to allow patients to continue the study treatment.
Dose intensity of study drugs | From first dose until study ends, approximately 4 years
  Dose intensity is computed as the ratio of actual cumulative dose received to actual duration of exposure.
ORR2 | Every 8-12 weeks until study ends, approximately 4 years
  Modified objective response rate (ORR2) per RECIST v1.1 (taking as baseline the most recent assessment prior to initiating combination)

SECONDARY OUTCOMES:
ORR | Every 8-12 weeks until study ends, approximately 4 years
  Overall response rate (ORR) per RECIST v1.1
PFS | Every 8-12 weeks until study ends, approximately 4 years
  Time from the date of first dose of study treatment to the date of first documented disease progression (per RECIST v1.1) or death due to any cause
DCR | Every 8-12 weeks until study ends, approximately 4 years
  Proportion of patients with best overall response of CR, PR, or SD
DOR | Every 8-12 weeks until study ends, approximately 4 years
  Time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause
Time to response | Every 8-12 weeks until study ends, approximately 4 years
  Time to response is the time between start of treatment until first documented response per RECIST v1.1.
Area under the plasma concentration-time curve (AUC) of study drugs | From pre-dose up to 8 hours post-dose on Day 15 of Cycle 1. One cycle=28 days.
  Pharmacokinetic (PK) parameters calculated based on the plasma concentrations versus time profiles by using non-compartmental methods.
Maximum observed plasma concentration (Cmax) of study drugs | From pre-dose up to 8 hours post-dose on Day 15 of Cycle 1. One cycle=28 days.
  PK parameters calculated based on the plasma concentrations versus time profiles by using non-compartmental methods.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis
Locations (10):
- Novartis Investigative Site, Toronto, Ontario, Canada
- Germany (2):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (3):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Singapore, Singapore
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: No